CLINICAL TRIAL: NCT03438994
Title: Toward Early Autism Assessment: A Prospective Diagnostic Accuracy Study
Brief Title: Early Assessment of Autism Through Smart Tablet Gameplay
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Strathclyde (Other)
Collaborators: Harimata (Unknown); University of Glasgow (Other); University of Aberdeen (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Jonathan Delafield-Butt, Principal Investigator, Director Laboratory for Innovation in Autism, University of Strathclyde
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: UEC17/49
Record Dates: First submitted 2018-02-10; First posted 2018-02-20 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Autism Spectrum Disorder; Other Neurodevelopmental Disorder
Keywords: autism; movement; tablet; gameplay
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This study will follow the "Standard for Reporting Diagnostic accuracy studies" (STARD) guidelines
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Participants diagnosed with ASD (Active Comparator)
  Interventions: Diagnostic Test: Play.Care
- Participants diagnosed with OND (Experimental)
  Interventions: Diagnostic Test: Play.Care
- Typically developing participants (Active Comparator)
  Interventions: Diagnostic Test: Play.Care

INTERVENTIONS:
Diagnostic Test: Play.Care — iPad based game to assess movement as the player interacts with the screen

SUMMARY:
The primary aim of this study is to compare the diagnostic accuracy of an iPad application (Play.Care assessment) with the current clinical "gold standard" diagnosis for diagnosis of Autism Spectrum Disorder (ASD) in children. Recent evidence has suggested that movement abnormalities are one of the early markers of ASD. However, current clinical diagnostic assessments fail to take this into account. Further, the current "gold standard" clinical tests take a number of hours to administer, require extensive clinical training and are subject to a certain level of subjectivity. Alternatively, by assessing a child's interaction with an iPad screen as they play, an objective measurement of movement can be obtained, which can aid in the diagnostic process.

This study aims to recruit a total of 760 children (Typically Developing (TD), Other Neurodevelopmental Disorders (OND) and ASD groups) to assess the diagnostic accuracy of tablet game play in ASD. Children who have been diagnosed with ASD will perform the Play.Care assessment to assess if the tablet result matches their clinical diagnosis. Results from the clinical assessment and Play.Care assessment will then be compared to assess the sensitivity (the proportion of participants with ASD who test positive for ASD as a result of the Play.Care assessment) and specificity (the proportion of participants without ASD who test negatively for ASD as a result of the Play.Care assessment assessment) of the Play.Care assessment.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) has, historically, been described as primarily a socio-cognitive disorder. While it has been noted that individuals with ASD may exhibit movement abnormalities such as altered gait or increased clumsiness, recent evidence has suggested the possible presence of an underlying motor disruption, common to individuals with ASD. By using smart tablet technology with built in 3 dimensional gyroscopes and accelerometers, we are now able to assess the movement of children with ASD as they interact with tablet screens during game play. It is proposed that this could be an enlightening avenue for assessment or even diagnosis of ASD.

The primary aim of this study is to clinically validate the ability of a new iPad game (called Play.Care) for diagnosis of ASD in children aged 30 months to 5 years (inclusive).

Three groups of participants will be recruited: children with a clinical diagnosis of ASD, children with a clinical diagnosis of an Other Neurodevelopmental Disorder (OND) and children developing typically (TD). A total of 760 children will be recruited between two cities, Glasgow, Scotland, United Kingdom and Gothenburg, Sweden. Gothenburgh will recruit 180 participants diagnosed with ASD, 60 participants diagnosed with OND and 100 typically developing participants. Glasgow will recruit 100 participants diagnosed with ASD, 140 participants diagnosed with OND and 180 participants developing typically.

Children developing typically will be recruited from local private nurseries. Children diagnosed with ASD or OND will be recruited from clinical diagnostic centres and specialist or inclusive schools.

Parents of children will be given a Participant Information Sheet and sign a Consent Form under protocol approved by health services (Glasgow and Gothenburg) and University ethics committees.

If the family is happy to participate, the child can either complete the Play.Care game in the clinic, during preschool hours in the preschool, or, if it is more suitable for the family, the researcher can come to their home. In either case, at the start of the data collection appointment, the parents must sign the consent form. Further information about the child's emotional state on the day of data collection will be recorded (e.g. mood, arousal, cooperativity). If the parents consented to their child being video recorded, a video camera will be setup prior to game play. This will give more information about the overall movement of the child as they play. The iPad will then be introduced to the child. Two games will be played. The first game is called 'Sharing' and requires the child to tap a piece of food to split it into 4 pieces and share it amongst game characters. The second game is called 'Creativity' and requires the child to choose an animal or object to trace and colour in. Each game has a two minute training phase followed by a five minute assessment phase. While the child is playing the games, or at an appropriate time, parents will be asked to complete 3 questionnaires about their child's everyday behaviour. These are standard assessments for children with ASD or OND and will help us understand how the information from Play.Care relates to everyday behaviour. These are the Strengths and Difficulties Questionnaire (SDQ), the Early Symptomatic Syndromes Eliciting Neurodevelopmental Clinical Examinations Questionnaire (ESSENCE-Q) and the Adaptive Behaviour Assessment Scale (ABAS). In some cases, information gathered during normal clinical assessment will also be gathered, namely but not exclusively the Vinelands Adaptive Behaviour Scale (VABS) and the Wechsler Preschool & Primary Scale of Intelligence (WPPSI). Once the questionnaires and the Play.Care assessment are complete, no further participation is required.

ELIGIBILITY:
1. Inclusion Criteria:

   1. All participants:

      * Aged 30 months - 5 years inclusive
   2. ASD Participants:

      * Diagnosis of autism spectrum disorder on the basis of DSM-V criteria or equivalent ICD-10 framework (F84): childhood autism (F84.0), atypical autism (F84.1), and Asperger's syndrome (F84.5)
   3. OND participants:

      * Other childhood developmental disorders including, but not limited to,
      * Attention Deficit Hyperactivity Disorder,
      * Developmental Coordination Disorder,
      * Intellectual disability,
      * Non- verbal disability and
      * Communication Disability.
      * Sensory and motor impairments will be included
2. Exclusion Criteria:

   1. Typically developing participants:

      * Diagnosis or suspicion of
      * Neuropathology
      * Psychopathology
      * Sensory or motor disorder including mild tremors
   2. ASD participants:

      * Uncorrected sensory (visual, hearing) impairments
      * Presence of any motor impairments or behavioural impairment that may obstruct testing
   3. OND participants:

      * Sub-clinical or secondary expressions of ASD
      * Uncorrected hearing or vision impairments

Ages: 30 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 760 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of Play.Care to detect ASD | Single data collection time point of 15 minutes for each subject.
  sensitivity and specificity of Play.Care to detect ASD

SECONDARY OUTCOMES:
Ability of Play.Care to distinguish ASD from OND | Single data collection time point of 15 minutes for each subject.
  sensitivity and specificity of Play.Care to distinguish ASD from OND

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Delafield-Butt, PhD, Principal Investigator — jonathan.delafield-butt@strath.ac.uk
Locations (2):
- Gillberg Neuropsychiatry Centre, Gothenburg, Sweden
- University of Strathclyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Millar L, McConnachie A, Minnis H, Wilson P, Thompson L, Anzulewicz A, Sobota K, Rowe P, Gillberg C, Delafield-Butt J. Phase 3 diagnostic evaluation of a smart tablet serious game to identify autism in 760 children 3-5 years old in Sweden and the United Kingdom. BMJ Open. 2019 Jul 16;9(7):e026226. doi: 10.1136/bmjopen-2018-026226. PMID 31315858